CLINICAL TRIAL: NCT00499694
Title: Phase II Trial of Bevacizumab and Satraplatin in Docetaxel Treated Metastatic Androgen Independent Prostate Cancer
Brief Title: Satraplatin and Bevacizumab in Treating Patients With Metastatic Prostate Cancer Previously Treated With Docetaxel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ulka Vaishampayan, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000518085; P30CA022453 (NIH); WSU-2006-118 (Other: Barbara Ann Karmanos Cancer Institute)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; satraplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Satraplatin (Experimental): Bevacizumab 10mg/kg,Intravenous, Day 1 of each Cycle (every 35 days) 15mg/kg,Intravenous, Day 15 of each Cycle (every 35 days)
  Satraplatin 80 mg/m(2), Orally, Days 1-5, every 35 days
  Interventions: Biological: bevacizumab; Drug: satraplatin

INTERVENTIONS:
Biological: bevacizumab — 10mg/kg,Intravenous, Day 1 of each Cycle (every 35 days) 15mg/kg,Intravenous, Day 15 of each Cycle (every 35 days)
  Other Names: Avastin ®
Drug: satraplatin — 80 mg/m(2), Orally, Days 1-5, every 35 days

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as satraplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving satraplatin together with bevacizumab may kill more tumor cells.

PURPOSE: This clinical trial is studying how well giving satraplatin together with bevacizumab works in treating patients with metastatic prostate cancer previously treated with docetaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with metastatic androgen-independent prostate cancer previously treated with docetaxel currently treated with satraplatin and bevacizumab.

Secondary

* Determine the toxicity of this regimen in these patients.
* Assess the prostate-specific antigen (PSA) response rate in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Assess changes in levels of N-terminal collagen peptide (NTX) and bone-specific alkaline phosphatase (BSAP) in patients treated with this regimen.
* Correlate urine NTX and serum BSAP levels with time to progression in patients treated with this regimen.

OUTLINE: Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral satraplatin on days 1-5. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 28-42 days.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate, meeting the following criteria:

  * Metastatic disease
  * Objective progression or rising prostate-specific antigen (PSA) despite androgen-deprivation therapy and antiandrogen withdrawal
* Patients with rising PSA must demonstrate a rising trend with 2 successive elevations at a minimum interval of 1 week

  * Minimum PSA of 5 ng/mL or new areas of bony metastases on bone scan required if no measurable disease
  * No minimum PSA for measurable disease
* Must have received ≤ 1 prior docetaxel-based chemotherapy for metastatic disease
* No known CNS disease or brain metastases
* Testosterone < 0.5 ng/mL (castrate level)

  * Concurrent luteinizing-hormone releasing-hormone agonist allowed to maintain castrate level

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin normal
* Creatinine ≤ 2 mg/dL OR creatinine clearance ≥ 50 mL/min
* Urine protein:creatinine ratio ≤ 1.0 OR proteinuria ≤ 2+ by urine dipstick OR ≤ 1 g protein/24-hour urine collection
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No significant traumatic injury within the past 28 days
* Adequately controlled hypertension (defined as systolic blood pressure [BP] ≤ 150 mm Hg and/or diastolic BP ≤ 100 mm Hg on antihypertensive medications)
* No history of hypertensive crisis or hypertensive encephalopathy
* No New York Heart Association class II-IV congestive heart failure
* No myocardial infarction or unstable angina within the past 6 months
* No stroke or transient ischemic attack within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* No symptomatic peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No prior malignancy except adequately treated skin cancer or any other cancer in complete remission for ≥ 2 years
* Able to swallow and retain capsules
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious nonhealing wound, ulcer, or bone fracture
* No known hypersensitivity to any component of bevacizumab
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to bevacizumab
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric illness or social situation that would preclude compliance with study requirements
* No HIV positivity
* No immune deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior flutamide
* More than 6 weeks since prior bicalutamide or nilutamide
* At least 4 weeks since prior radiotherapy
* At least 2 weeks since prior minor surgery
* More than 7 days since prior core biopsy or minor surgery (excluding placement of a vascular access device)
* More than 28 days since prior major surgery or open biopsy (8 weeks if high-risk procedure such as liver resection, thoracotomy, or neurosurgery)
* Concurrent low-dose aspirin (≤ 325 mg/day) allowed
* Concurrent anticoagulants allowed if patient has been on therapy ≥ 4 weeks and has no acute thromboembolic activity
* No concurrent major surgery
* No concurrent aprepitant
* No concurrent immunosuppressive therapy
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent antitumor therapy (including radiotherapy)
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab and Satraplatin: Bevacizumab 10mg/kg,Intravenous, Day 1 of each Cycle (every 35 days) 15mg/kg,Intravenous, Day 15 of each Cycle (every 35 days)
  Satraplatin 80 mg/m(2), Orally, Days 1-5, every 35 days
  bevacizumab: 10mg/kg,Intravenous, Day 1 of each Cycle (every 35 days) 15mg/kg,Intravenous, Day 15 of each Cycle (every 35 days)
  satraplatin: 80 mg/m(2), Orally, Days 1-5, every 35 days
Period: Overall Study
Arm/Group | Bevacizumab and Satraplatin
Started | 31
Completed | 30
Not Completed | 1
Not completed — Patient never received treatment. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Satraplatin
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. TTP is measured using Kaplan-Meier product-limit.
Time Frame: Every 70 days
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Bevacizumab and Satraplatin: Bevacizumab: 10mg/kg,Intravenous, Day 1 of each Cycle (every 35 days) Bevacizumab: 15mg/kg,Intravenous, Day 15 of each Cycle (every 35 days)
  Satraplatin: 80 mg/m(2), Orally, Days 1-5, every 35 days
Arm/Group | Bevacizumab and Satraplatin
Number analyzed (Participants) | 31
months | 7.0 [4.7 to 8.5]

2. Secondary Outcome: Toxicity, Presented as the Number of Participants With Adverse Events
Description: Toxicity was categorized according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (version 3.0).
Time Frame: Day 1 of every cycle (35 days) and Day 15 of every cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and Satraplatin
Number analyzed (Participants) | 31
Participants
  Nausea | 16
  Vomiting | 11
  Diarrhea | 10
  Leukopenia | 14
  Neutropenia | 10
  Anemia | 12
  Edema | 3
  Dehydration | 8
  Hyperglycemia | 21
  Thrombocytopenia | 19
  Proteinuria | 18
  Hypertension | 4
  Fatigue | 19
  Hypokalemia | 5
  Hyponatremia | 5
  hypomagnesemia | 4
  AST | 7
  Creatinine | 1
  Constipation | 5
  Bloating/Distention | 2
  Fever/Rigors | 1
  Dyspepsia | 6
  Weight Loss | 7
  Anorexia | 8
  Allergic Reaction | 2

3. Secondary Outcome: Percentage of Participants With Prostate-specific Antigen (PSA) Response
Description: Prostate-specific antigen (PSA) response rate as measured by a 50% or better decrease in PSA levels
Time Frame: Day 1 of every cycle (35 days) and Day 15 of every cycle
Measure: Number (90% Confidence Interval); unit: pct. of pts. with 50%+ decrease in PSA
Arm/Group | Bevacizumab and Satraplatin
Number analyzed (Participants) | 30
pct. of pts. with 50%+ decrease in PSA | 17 [8 to 30]

4. Secondary Outcome: Overall Survival
Description: Overall survival using the Kaplan-Meier method
Time Frame: Followed every 3 months after treatment is discontinued
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bevacizumab and Satraplatin
Number analyzed (Participants) | 31
months | 11.2 [9.1 to 16.4]

ADVERSE EVENTS:
Arm/Group | Bevacizumab and Satraplatin
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Satraplatin (N=30)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Leukeopenia (Investigations) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Fatigue (Gastrointestinal disorders) | 1 (1)
Thrombosis_PE (Vascular disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Bloating Distention (Gastrointestinal disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Satraplatin (N=30)
Nausea (Gastrointestinal disorders) | 16 (16)
Vomiting (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Leukopenia (Blood and lymphatic system disorders) | 14 (14)
Neutropenia (Blood and lymphatic system disorders) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Edema (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 8 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (19)
Proteinuria (Renal and urinary disorders) | 18 (18)
Hypotension (Vascular disorders) | 4 (4)
Fatigue (General disorders) | 19 (19)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
AST (Investigations) | 7 (7)
Creatinine (Investigations) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (5)
Bloating Distention (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Weight loss (Investigations) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Allergic Reaction (Immune system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size, correlative ERCC testing conducted in only a subset of patients (14 of 30 pts) and the findings of this study are hypothesis generating however validation in larger sample size would be needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes